CLINICAL TRIAL: NCT06912347
Title: Acupoint Application Combined With Herbal Fumigation and Wash for Preventing Diarrhea-induced Perianal Infection in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation:A Single-Center, Randomized, Controlled, Open-Label Clinical Study
Brief Title: Acupoint Application With Herbal Fumigation and Wash for Preventing Diarrhea-induced Perianal Infection in Allo-HSCT Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Xiaoxia, Prof, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025125
Record Dates: First submitted 2025-03-24; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupoint Application Combined With Herbal Fumigation and Wash Group (Experimental): Starting 24 hours before pre-treatment, the participants will receive herbal fumigation of the perianal area twice daily (morning and afternoon), with each session lasting 5 minutes. Additionally, starting 30 minutes after each meal, acupoint application will be performed on five acupoints: Shenque (CV8), Tianshu (ST25), and bilateral Zusanli (ST36). The application will last 4 hours per day.
  Interventions: Other: Intervention Group
- Povidone-iodine warm water fumigation Group (Active Comparator): Starting 24 hours before pre-treatment, the participants will receive povidone-iodine warm water fumigation of the perianal area twice daily (morning and afternoon), with each session lasting 15 minutes.
  Interventions: Other: control group

INTERVENTIONS:
Other: Intervention Group — Starting 24 hours before pre-treatment, you will receive herbal fumigation of the perianal area twice daily (morning and afternoon), with each session lasting 5 minutes. Additionally, starting 30 minutes after each meal, acupoint application will be performed on five acupoints: Shenque (CV8), Tianshu (ST25), and bilateral Zusanli (ST36). The application will last 4 hours per day.
  Arms: Acupoint Application Combined With Herbal Fumigation and Wash Group
Other: control group — Starting 24 hours before pre-treatment, you will receive povidone-iodine warm water fumigation of the perianal area twice daily (morning and afternoon), with each session lasting 15 minutes.
  Arms: Povidone-iodine warm water fumigation Group

SUMMARY:
The goal of this clinical trial is to evaluate whether the combination of herbal fumigation and acupoint application can effectively prevent diarrhea in patients undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT).The main questions it aims to answer are:

Does the combination of herbal fumigation and acupoint application reduce the incidence of diarrhea in allo-HSCT patients? Does this intervention improve patients' quality of life and reduce the risk of perianal infections? Researchers will compare the intervention group (herbal fumigation + acupoint application) to the control group (povidone-iodine warm water fumigation) to determine the effectiveness of the TCM-based approach in preventing diarrhea and related complications.

Participants will:

Receive either herbal fumigation and acupoint application or povidone-iodine warm water fumigation twice daily, starting from 24h before transplant conditioning until 30 days post-transplantation (Day +30).

Undergo daily monitoring of perianal and local skin conditions, as well as diarrhea symptoms, by trained professionals.

This study aims to provide evidence for a non-invasive, low-risk TCM approach to improving outcomes for allo-HSCT patients.

DETAILED DESCRIPTION:
Diarrhea is one of the most common complications following hematopoietic stem cell transplantation (HSCT), with an incidence rate of 50%-70%. During HSCT, high-dose chemotherapy drugs can damage the intestinal mucosa, especially in allogeneic haploidentical hematopoietic stem cell transplantation, where the pre-treatment dosage is 5-10 times higher than that of conventional chemotherapy. This makes patients prone to chemotherapy-related diarrhea. Additionally, due to the patients' compromised immune systems, they are susceptible to other related types of diarrhea. Prolonged diarrhea can easily lead to damage to the perianal skin and intestinal mucosa, severely affecting the quality of life while increasing the risk of perianal infections. This, in turn, may trigger severe systemic infections, sepsis, organ failure, and ultimately transplant failure. Currently, the main causes of diarrhea are believed to include chemotherapy toxicity, infections, acute graft-versus-host disease (aGVHD), engraftment syndrome, and thrombotic microangiopathy. Chemotherapy-related diarrhea is most common in the early stages of transplantation, with an incidence rate of 78.5%, and a median onset time of -3 days (range: -9 to +10 days). The clinical manifestations of diarrhea are complex, and the mortality rate is high, with some studies reporting rates as high as 38.7%. Effectively preventing diarrhea is of great significance for improving patients' quality of life and prognosis.

In Western medicine, the management of diarrhea primarily focuses on symptom control, promoting mucosal repair, preventing secondary infections, and maintaining water and electrolyte balance. While these approaches have achieved certain clinical efficacy, they still have limitations, particularly in the prevention of diarrhea. Traditional Chinese medicine (TCM), characterized by its principles of "syndrome differentiation and treatment" and a "holistic approach," offers greater flexibility. With ongoing research, the efficacy of TCM in treating diarrhea has gradually become evident. Previous studies have shown that the mechanisms of TCM in alleviating diarrhea in chemotherapy patients include: increasing colonic cyclooxygenase-2 and prostaglandin B2 levels, reducing the movement of water and electrolytes into the intestinal lumen; promoting the production of serum IL-15, increasing cecal pH, reducing colonic β-glucuronidase activity, and protecting the structural integrity of the intestinal mucosa; promoting the secretion of intestinal IgA, increasing the content of vasoactive intestinal peptide, reducing pro-inflammatory factors such as IL-15, and regulating intestinal immune barrier function.

Herbal fumigation and external application are important components of TCM external therapies. Warm liquids can promote blood circulation, working synergistically with herbal medicine to unblock qi and blood, dredge meridians, and dispel cold and pain. High concentrations of active drug components act locally on the body, while also avoiding the metabolic burden on the liver and kidneys associated with oral administration of herbal medicine. With minimal side effects, these methods are worthy of clinical promotion. This study aims to explore the clinical application of herbal fumigation and acupoint application in preventing diarrhea in HSCT patients, with the goal of reducing the incidence of diarrhea and improving patients' quality of life and prognosis.

If the participant agree to participate in this study, he/she will be randomly assigned to either the intervention group or the control group, with an equal probability of being placed in either group. Each group will include 90 participants.

* Intervention Group: Starting 24 hours before pre-treatment, the participants will receive herbal fumigation of the perianal area twice daily (morning and afternoon), with each session lasting 5 minutes. Additionally, starting 30 minutes after each meal, acupoint application will be performed on five acupoints: Shenque (CV8), Tianshu (ST25), and bilateral Zusanli (ST36). The application will last 4 hours per day.
* Control Group: Starting 24 hours before pre-treatment, the participants will receive povidone-iodine warm water fumigation of the perianal area twice daily (morning and afternoon), with each session lasting 15 minutes.

After enrollment, the participants will be assigned a unique identification number, and a medical record will be created for them. During the study,the participants will be required to cooperate with the research team in implementing the assigned perianal care measures. The research team will observe and record their daily perianal and local skin conditions, as well as any occurrences of diarrhea. All interventions will be performed and monitored by trained professionals.

All information will be managed by the project contact person (Qin Liyuan) and will only be accessible to members of the research team. It will not be shared with individuals outside the research team. If any remaining data is to be used for future research after the study concludes, it will only be used with the participants' consent.

By participating in this study, the participants will receive either herbal fumigation and acupoint application or standard perianal care, depending on your group assignment. The research team will closely monitor the participants' health status, aiming to reduce the incidence of diarrhea and improve prognosis.

ELIGIBILITY:
Inclusion Criteria:

* First-time recipient of allogeneic hematopoietic stem cell transplantation.
* Age between 14 and 70 years old, regardless of gender.
* Primary disease type: Hematologic malignancies or aplastic anemia, with no restrictions on disease stage or remission status.
* Transplant type: Matched sibling donor, haploidentical related donor, or unrelated donor.
* Transplant conditioning regimen: Myeloablative, reduced-intensity, or non-myeloablative.
* Informed consent and voluntary participation in this clinical study.

Exclusion Criteria:

* Presence of intestinal infection within 2 weeks prior to enrollment.
* Previous diagnosis of inflammatory bowel disease or irritable bowel syndrome.
* Pathologically or radiologically confirmed involvement of the primary disease in the intestines.
* ECOG performance status ≥ 2, or presence of organ failure, rendering the patient unable to tolerate allogeneic hematopoietic stem cell transplantation.
* Allergy to the trial medications or physical conditions unsuitable for sitz baths.
* Individuals with mental disorders or those unable to provide informed consent.
* Poor compliance, such as failure to implement the intervention measures for 3 consecutive days.
* HIV-infected individuals, or those with a history of drug abuse or chronic alcoholism that may affect the evaluation of trial results.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-03-18 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who suffered from different diarrhea severity | From the beginning of pretreatment to 30 days after transplantation
  The severity of diarrhea was assessed using the ECOG version of the Common Toxicity Criteria (CTC) grading system:
  Grade 0: No diarrhea Grade 1: 2-3 loose stools per day above baseline Grade 2: 4-6 loose stools per day above baseline Grade 3: 7-9 loose stools per day above baseline Grade 4: ≥10 loose stools per day above baseline with dehydration or requiring parenteral nutrition (Severe diarrhea was defined as ≥Grade 3)
Number of participants who suffered from perianal infection | From the beginning of pretreatment to 30 days after transplantation
  Perianal Infection Grading adapted from WHO guidelines for perianal infection assessment:
  Grade 0 (No infection): Intact perianal skin/mucosa, dry and clean, asymptomatic Grade 1: Induration and/or mucosal erythema, painful defecation without bleeding Grade 2: Perianal erythema with swelling/tenderness, OR skin fissures <0.5cm Grade 3: Abscess formation OR fissures ≥0.5cm with surrounding inflammation

SECONDARY OUTCOMES:
Number of participants who suffered from different hemorrhoids Grade | From the beginning of pretreatment to 30 days after transplantation
  Hemorrhoid Grading according to the Goligher Classification:
  Grade I: Rectal bleeding (dripping or jet-like) during defecation, self-limiting; no prolapse Grade II: Recurrent bleeding; prolapse during defecation with spontaneous reduction Grade III: Occasional bleeding; prolapse requiring manual reduction (induced by defecation, exertion, or prolonged standing) Grade IV: Persistent prolapse (irreducible or immediately recurrent) with potential complications (infection, edema, erosion, necrosis, severe pain)
Number of participants who suffered from acute intestinal graft-versus-host disease | From the beginning of pretreatment to 100 days after transplantation
  acute Graft-versus-Host Disease (aGVHD) of the Gut: Diagnostic Criteria:
  ≥3 loose stools/day (total volume ≥500mL/day in adults) Exclusion of infectious/medication-related causes, conditioning toxicity, and transplant-associated microangiopathy Endoscopic findings: Colorectal edema/ulceration (most common)
Number of participants who suffered from non-recurrent death | From the beginning of pretreatment to 100 days after transplantation
  Non-Relapse Mortality (NRM): Death unrelated to primary disease recurrence, typically including:
  Infection (bacterial/viral/fungal) Graft-versus-host disease (GVHD) Organ toxicity (e.g., hepatic/renal/pulmonary) Transplant-related complications (e.g., hemorrhage, VOD/SOS) Secondary malignancies

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD Sharing Time Frame: Starting 6 months after publication, available for 5 years.
Access Criteria: De-identified IPD will be shared with qualified researchers who provide a methodologically sound proposal. Data requests should include:
  Specific analysis objectives Statistical methods plan Ethics approval proof
  Approved requestors will gain access to:
  Anonymized participant-level data Study protocol/SAP Analytical codebook
  Access process:
  Submit proposal to [qly02Q05@rjh.com.cn] Institutional review (4-week turn around) Data transfer via encrypted platform after DUA execution